CLINICAL TRIAL: NCT02196662
Title: Pharmacokinetics of IBD98-M 400mg-57.5/Day in Healthy Volunteers
Acronym: IBD98-M
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Holy Stone Healthcare Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 110200
Record Dates: First submitted 2014-07-15; First posted 2014-07-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment A (Experimental): IBD98-M: mesalamine-sodium hyaluronate 200mg-28.75mg X2
  Interventions: Drug: IBD98-M:
- Treatment B (Experimental): IBD98-M without HA: Mesalamine 200mg X2
  Interventions: Drug: IBD98-M without HA
- Treatment C (Experimental): Delzicol 200 mg X2
  Interventions: Drug: Delzicol

INTERVENTIONS:
Drug: IBD98-M: — single adiministration
  Other Names: Mesalamine-Sodium Hyaluronic 400 mg-57.5 mg
  Arms: Treatment A
Drug: IBD98-M without HA — single adiministration
  Other Names: IBD98-M without HA: Mesalamine 400 mg
  Arms: Treatment B
Drug: Delzicol — single adiministration
  Other Names: Mesalamine 400 mg
  Arms: Treatment C

SUMMARY:
The primary objective of this study is to compare the rate and extent of absorption of mesalamine-sodium hyaluronate 200 mg-28.75 mg delayed-release capsule (IBD98-M, Test) versus Delzicol 400 mg delayed-release capsule (mesalamine Reference), administered as a single oral dose of 2 x 200 mg-28.75 mg delayed-release capsule (total dose of 400 mg-57.50 mg) or 1 x 400 mg delayed-release capsule under fasting conditions.

DETAILED DESCRIPTION:
Safety population The safety population is defined as all subjects who received at least one dose of the study medication.

Pharmacokinetic Population The pharmacokinetic population will include all subjects completing at least 2 periods and for whom the pharmacokinetic profile can be adequately characterised.

Any subject with pre-dose concentrations for mesalamine will be excluded from the pharmacokinetic population for this analyte if the pre-dose concentration is greater than 5% of the Cmax value of that period for this subject.

Data from subjects who experienced emesis during the sampling interval and who were not withdrawn as per criterion established under section 9.10 may be evaluated after completion of the pharmacokinetic analysis. Any subject who experienced emesis within 2 times median Tmax of the current study (based on the Reference product) will be excluded from the statistical analysis. Data (concentrations and pharmacokinetic parameters) from subjects excluded due to a pre dose concentration greater than 5% of their Cmax or from subjects withdrawn due to adverse events or vomiting episodes will be presented but excluded from descriptive statistics.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, smoker (no more than 25 cigarettes daily) or non-smoker, 18 years of age and older, with BMI > 18.5 and < 30.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Healthy as defined by:

   * the absence of clinically significant illness and surgery within 4 weeks prior to dosing. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Qualified Investigator.
   * the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
   * the absence of history or known pyloric stenosis.
   * the absence of known gastric or duodenal ulcer.
   * the absence of urinary tract obstruction.
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive method throughout the study and for 30 days after the last study drug administration:

   * intra-uterine contraceptive device placed at least 4 weeks prior to study drug administration
   * condom with intravaginally applied spermicide starting at least 14 days prior to study drug administration
   * hormonal contraceptives starting at least 4 weeks prior to study drug administration and must agree to use the same hormonal contraceptive throughout the study
   * sterile male partner (vasectomized since at least 6 months).
4. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen at screening.
3. History of allergic reactions to mesalamine, salicylates, aminosalicylates, hyaluronic acid, or other related drugs.
4. Positive pregnancy test at screening.
5. Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
6. Clinically significant electrocardiogram (ECG) abnormalities or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
7. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
8. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to screening.
9. Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics) prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
10. Use of medication other than topical products without significant systemic absorption and hormonal contraceptives:

    * prescription medication within 14 days prior to the first dosing;
    * over-the-counter products including natural health products (e.g. food supplements and herbal supplements) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    * a depot injection or an implant of any drug (other than hormonal contraceptives) within 3 months prior to the first dosing.
11. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
12. Hemoglobin <128 g/L (males) and <115 g/L (females) and hematocrit <0.37 L/L (males) and <0.32 L/L (females) at screening.
13. Breast-feeding subject.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve in plasma of IBD98-M | Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Denis Audet, M.D., Principal Investigator — inVentiv
Locations (1):
- inVentiv Health Clinique, Québec, Quebec, Canada